CLINICAL TRIAL: NCT03446014
Title: The Genetic and Risk Factor Contribution to the Progression of Peripheral Artery Disease and Severe Adverse Events
Brief Title: PAD Registry and Fitbit Sub-Study Program
Acronym: PADR
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 817194
Record Dates: First submitted 2015-07-21; First posted 2018-02-26 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group for Fitbit Sub-Study: Patient will be given Fitbit device, but will have no access to Fitbit website or interface. The coordinator will set up the patient's Fitbit on the office computer and will have access to the fitbit's associated username and password (this will be generated by the coordinator). The patient will be instructed to walk as much as they can each day, and to check the Fitbit wrist band periodically throughout the day to view their walking progress. At the end of the three month intervention, the patient will complete questionnaires and undergo a repeat 6 minute walk test.
  Interventions: Device: Fitbit Sub-Study
- Intervention Group for Fitbit Sub-Study: Patient will be given the Fitbit device and instructed on how to use it. They will be given their username and password to the Fitbit device, and instructed on how to interact with other patients in the study as well as the coordinator on the Fitbit website. The coordinator will also show the patient how to install the application on a smart phone device and use the device via smartphone. The patient will then be instructed to walk as far as they can each day for a period of 12 weeks. Patients will check their steps daily and interact with other patients who participate in the study. Patients will return for a 3 month follow-up appointment where they will undergo a redo 6 minute walk test and questionnaires.
  Interventions: Device: Fitbit Sub-Study

INTERVENTIONS:
Device: Fitbit Sub-Study

SUMMARY:
The genetic contribution and influence on the progression of peripheral artery disease (PAD) and possible cardiovascular events remains relatively unknown. As a result, the investigators are proposing for the creation of a registry of patients in the University of Pennsylvania Health System who are known to have PAD. The patients in this registry will be systematically monitored by conducting lower extremity ultrasound exams, ankle-brachial index (ABI) measurements, and six minute walk tests which have strong value in the positive diagnoses of PAD. These exams, combined with follow-up quality of life questionnaires, would allow for thorough monitoring of new diagnoses, symptoms, or serious adverse events. Blood will also be drawn looking for genetic biomarkers associated with this disease, which will provide further knowledge on the advancement and potential cardiovascular events associated with this disease. This blood will also be analyzed for components that will provide the investigators with knowledge of the patients overall blood vessel health. Micro RNA will also be evaluated to try to test if proteins and RNA in the blood can be used as predictors for future strokes or heart attacks. These exams will be repeated once annually over a duration of 10 years, with patients having hemodynamic monitoring as well as quality-of-life and cardiovascular events recorded at each visit. The data obtained from this registry will be compared to a created genetic profile looking for any genetic contribution to these new developments. Furthermore, this knowledge should offer impetus for physicians to target patients with these risk factors for the identification of potential adjustments to care.

DETAILED DESCRIPTION:
500 subjects will be recruited from the general Philadelphia community and from the University of Pennsylvania Healthcare System. This population will be carefully characterized with assessment for cardiovascular risk factors to include smoking, diabetes mellitus, hypertension, and previous surgery or vascular interventions. Those patients with the presence of diabetes, hypertension, and hypercholesterolemia will be considered positive if they are being prescribed drugs for each respective condition. Physician's clinics will be screened for patients who meet the necessary inclusion criteria. These physicians will then be contacted for permission to speak with the patient. Upon approval, a coordinator will contact the patient regarding the study and to gauge interest. If interested, the coordinator will go through a screening form with the patient, as well as schedule a baseline visit. Subjects will also be recruited from Upenn research database comprised of subjects who have participated in previous research studies and who have asked to be contacted for future studies, such as CVI BioBank, Genetics of Cardiovascular and Metabolic Phenotypes (IRB #808346). Potential subjects will also be recruited via Penn Data Store. Patients who cannot be contacted directly will be contacted through the mail.

For their baseline visit, patients will be asked to read and sign the consent form, as well as approached for participation in the CVI BioBank, Genetics of Cardiovascular and Metabolic Phenotypes (IRB# 808346). Additionally, patients will be given the option of participating in the activity monitoring sub-study. Patients will then asked to undergo an ABI measurement using standardized methods - brachial and ankle systolic pressures will be measured with appropriately sized cuffs attached to sphygmomanometers. Return of flow will be determined using a continuous wave Doppler. In addition, patients will undergo a lower extremity duplex ultrasound evaluation of their arterial system, with plaque being used as a measure of disease progression. The evaluation will be done in coordination with the Inter-societal Commission for Accreditation of Vascular Laboratory Guidelines. In each follow-up exam, PAD progression will be defined as either a new stenosis or progression of a baseline stenosis to an occlusion. Furthermore, patients will undergo a 6-MWD test, with the primary unit of analysis being the total distance walked (in meters) regardless of whether the subjects stopped or not during the conduct of the test. Patients will also have 10 mLs of blood drawn, which will be evaluated for any genetic and vascular biomarkers that may have contributed to the disease (see Section 3.0 for Analysis and Evaluation). Micro RNA will also be evaluated for any predictors of future strokes or heart attacks. Study visits will be completed once annually over duration of 10 years, with questionnaires being repeated every 6 months via telephone. These questionnaires, the Walking Impairment Questionnaire (WIQ) and RAND-Item short Form Survey, will be completed and will ask the patients about any interval changes in medical history, any severe adverse events that may have occurred, and their overall quality of life.

Patients enrolled in the optional activity monitoring sub study will be randomized to one of two groups: intervention group or control group. Intervention group participants will receive an activity monitor device (Fitbit http://www.fitbit.com/) and instructed on its use. Additionally, coordinators will monitor the intervention groups usage of the device and make routine recommendations on their activity level using the Way To Health platform. Way to Health is an integrated research platform that uses online tools, wireless technologies, and other applications to allow investigators to test ways of improving health behaviors and helping people keep on track to better health. Patients in the intervention group will also receive financial incentives for wearing the Fitbit and also be entered into a lottery if they are reaching their goals. Patient's will be increased by the Way To Health program according to the algorithm described below:

* <5000 steps: 50% increase on goal
* 5,001 - 7,500 steps: 40% increase on goal
* 7,501 - 10,000 steps: 30% increase on goal ->10,000 steps: 20% increase on goal

Participants in the control group will receive an activity monitoring device that they will not be able to engage with but instructed to wear for monitoring purposes once a week every month. Each subject will perform the same procedures used on patients not enrolled in the sub-study. However, patients will be asked to return to our office for a 3 month follow-up visit for a repeat 6 minute walk test and Walking Impairment Questionairre (WIQ). The data recorded on the activity monitor device will be uploaded by the subjects for view via sync through proprietary software on a smartphone, tablet, or computer. The data will be password protected and will allow access to the investigator and the subjects randomized to the intervention group to have access.

ELIGIBILITY:
Inclusion Criteria:Patients between the ages of 18 and 90 and those patient's with PAD and other risk factors (smoking, diabetes mellitus, hypertension, and previous surgery or vascular interventions) will be included. These patients must have peripheral artery disease with objective vascular laboratory measurements that confirm disease. Moreover, patients will also be considered who have a history of PAD and a normal ABI after revascularizations. Patients will also be screened for any prior adverse events such as myocardial infarction or stroke.

Exclusion Criteria: Patients below that age of 18 and over the age of 90 who do not have a positive diagnosis or history of PAD will be excluded from the study. Pregnant and lactating women and those people unable to provide informed consent will also be excluded. A patient will have the option to not participate in the study and not sign the informed consent. If a patient declines to participate, there is no effect on the patient's regular, ongoing cardiac care. Patients who do not access to a smartphone/tablet/computer or cannot engage in active participation via the software program will be excluded from the Fitbit sub-study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Peripheral Artery Disease is a disease that is highly prevalent within the United States, affecting close to 8-12 million individuals. These individuals' qualities of life are likely impaired due to limited walking ability, shortness of breath, and claudication. In addition, it is well known that risk factors such as smoking, diabetes mellitus, hypertension, and dyslipidemia can play a role in the onset of this disease
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Registry creation of patients with known PAD | 10 Years
  Patients will be recruited from the University of Pennsylvania Health System via surveying of physician's clinics and various databases. Appropriate clinical staff will be informed of this study and its requirements prior to a patient's enrollment. As a result, routine care or other medical procedures of the patient will not be interfered with.

SECONDARY OUTCOMES:
Patient walking distance | 1 Year
  Patients enrolled in the optional sub-study concerning the use of activity monitoring will be randomized into one of two groups. Those patients randomized into the intervention group, with close monitoring, will exhibit increased motivation for activity and walk farther on their follow-up visit. This will be demonstrated by an increased number of laps walked at their 3 month follow-up visit. Additionally, these subjects would also exhibit increased flow as determined by their ultrasound at their yearly follow-up visit. This would be a result of increased motivation and tolerance for exercise and activity.

OTHER OUTCOMES:
Genetic and Vascular Testing of Patients | 10 Years
  Analysis: After overnight fasting, each patient will donate approximately 10 mLs of venous blood. Blood draws will be done on all patients and will look for genetic and vascular biomarkers that could contribute to progression of the disease. As stated, we are not searching for any new genes in individuals, but rather genetic trends in a large population. Blood will be drawn in plastic, sodium citrate tubes used for microparticles. These tubes will be spun at 2,500g x 15 minutes at room temperature. Closely monitoring these trends will help us define genetic alterations that could lead to the progression of disease.
Systematically Monitoring Patients | 10 Years
  Following enrollment into the study, patients will be systematically monitored for the entirety of the study. As stated, this will be conducted by annual visits the patients will undergo. These visits, in coordination with the procedures associated with them, will allow us to properly evaluate the progression of disease in these patients. Moreover, the questionnaires that will be conducted at 6 month intervals will ask patients about their overall quality of life and adverse events that may have occurred in the interim period. In doing so, we will be able to systematically monitor the progression of peripheral artery disease longitudinally in a large population, allowing us to draw conclusions as to the onset and time frame of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Emile R Mohler, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States